CLINICAL TRIAL: NCT00716209
Title: Infrastructure for Developing Gastrointestinal Cancer Prognostic and Predictive Markers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Haematology-Oncology (Other)
Responsible Party: Sponsor-Investigator, Haematology-Oncology, Ross Andrew Soo, National University Hospital, Singapore
Organization: National University Hospital, Singapore (Other)
Other Study IDs: NUSIRB 04-116
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients with cancers of the gastrointestinal tract (eg. colorectal, gastric, pancreatic, esophageal)

SUMMARY:
The proposal seeks to establish:

* A comprehensive compilation (database) of clinical information comprising clinical, histopathological, treatment and follow-up characteristics of past and future gastrointestinal cancer (GIC) cases in Singapore that can be shared by investigators. The characteristics will include clinical (eg age, sex, stage), histopathological (eg. grade, type), treatment (eg. treatment status, regimens) and outcome data (eg. survival, toxicity) from medical records.
* A collection (bank) of corresponding frozen and fixed tissue, blood and processed samples (enriched blood mononuclear cells, protein, RNA, DNA, tissue arrays) in Singapore that can be shared by the investigators.
* A gastrointestinal cancer co-operative group (GCCG) of clinicians and scientists researching prognostic and predictive markers in GIC, which will benefit from the multi-disciplinary knowledge, information and samples of its members.
* To characterise genetic polymorphisms related to Gastrointestinal cancer chemotherapy treatment in controls (healthy volunteers)

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancers of the gastrointestinal tract (eg. colorectal, gastric, pancreatic, esophageal)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To examine associations between candidate markers and patient response, toxicity and other clinicopathological characteristics, standard descriptive statistics will be used, according to the variable type (e.g. continuous, discrete, parametric, non-parametric). Associations with patient outcome will be assessed by Kaplan Meier analysis and independence examined in multivariate models by Cox proportional hazard analysis. To discriminate prognostic and predictive significance, outcome associations of candidate markers will be examined with respect to the treatment status of cohorts as outlined in the "Introduction" and as performed previously.
Sampling Method: Non-Probability Sample
Dates: Start 2012-09; Primary Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Andrew Soo, MBBS, Principal Investigator — National University Hospital, Singapore; Alex Chang, Principal Investigator — Johns Hopkins Singapore International Medical Centre; Chung Yip Chan, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Soong R, Robbins PD, Dix BR, Grieu F, Lim B, Knowles S, Williams KE, Turbett GR, House AK, Iacopetta BJ. Concordance between p53 protein overexpression and gene mutation in a large series of common human carcinomas. Hum Pathol. 1996 Oct;27(10):1050-5. doi: 10.1016/s0046-8177(96)90282-8. PMID 8892589
- [Background] Soong R, Powell B, Elsaleh H, Gnanasampanthan G, Smith DR, Goh HS, Joseph D, Iacopetta B. Prognostic significance of TP53 gene mutation in 995 cases of colorectal carcinoma. Influence of tumour site, stage, adjuvant chemotherapy and type of mutation. Eur J Cancer. 2000 Oct;36(16):2053-60. doi: 10.1016/s0959-8049(00)00285-9. PMID 11044641
- [Background] Mattison LK, Soong R, Diasio RB. Implications of dihydropyrimidine dehydrogenase on 5-fluorouracil pharmacogenetics and pharmacogenomics. Pharmacogenomics. 2002 Jul;3(4):485-92. doi: 10.1517/14622416.3.4.485. PMID 12164772